CLINICAL TRIAL: NCT07032285
Title: Multicenter, Open-Label Phase II Trial of Cirtuvivint in Selected Advanced Soft-Tissue Sarcomas
Brief Title: Cirtuvivint in Selected Advanced Soft-Tissue Sarcomas
Acronym: CIRTUSARC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asociación Europea y Latinoamericana SELNET para la Investigación en Sarcomas (Other)
Collaborators: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SELNET 7-2; 2024-511987-10-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-19; First posted 2025-06-23 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Soft Tissue Sarcoma (STS)
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Crituvivint (Experimental): Cirtuvivint (SM08502) will be administered orally at 80 mg/day, 5 days on/2 days off.
  Cirtuvivint is supplied as tablets containing 10 mg or 50 mg of the active pharmaceutical ingredient (API).
  Cirtuvivint is taken with water once a day (on dosing days) at the same time every day.
  Doses will be taken without food (foo restriciton 1 hour before treatment and 2 hours afterdosing).
  Doses delayed by 12 hours will be considered missed and should not be taken. If vomiting occurs,the dose must not be retaken.
  Cirtuvivint is dosed in 28-day continuous cycles (28 days of treatment will beconsidered as one cycle) Treatment will continue until disease progression, unacceptable toxicity or investigator/patient decision
  Interventions: Drug: Cirtuvivint

INTERVENTIONS:
Drug: Cirtuvivint — Cirtuvivint (SM08502) will be administered orally at 80 mg/day, 5 days on/2 days off. Cirtuvivint is supplied as tablets containing 10 mg or 50 mg of the active pharmaceutical ingredient (API). Cirtuvivint is taken with water once a day (on dosing days) at the same time every day. Doses will be taken without food (foo restriciton 1 hour before treatment and 2 hours afterdosing). Doses delayed by 12 hours will be considered missed and should not be taken. If vomiting occurs,the dose must not be retaken. Cirtuvivint is dosed in 28-day continuous cycles (28 days of treatment will beconsidered as one cycle) Treatment will continue until disease progression, unacceptable toxicity or investigator/patient decision

SUMMARY:
The study is a Phase 2 clinical trial of the drug cirtuvivint as a second-line treatment for advanced soft tissue sarcomas. The study is being conducted in Spain and is expected to enroll approximately 25 patients in total. The primary objective of this Phase 2 study is to evaluate the efficacy of treatment with cirtuvivint.

Cirtuvivint is an anti-cancer medication developed by the U.S. company Biosplice Therapeutics, Inc. This drug is an inhibitor of the enzymes CLK1-4 and DYRK1-4 (molecules involved in the cell cycle) and is administered as oral tablets. This product is still under investigation and has not yet been approved in Europe.

ELIGIBILITY:
Inclusion criteria:

1. Patients must provide written informed consent prior to performance of any study-specific procedures and must be willing to comply with treatment and follow up. Informed consent must be obtained prior to the start of the screening process. Procedures conducted as part of the patient's routine clinical management (e.g., imaging tests), obtained prior to signature of informed consent may be used for screening or baseline purposes as long as these procedures are conducted as specified in the protocol.
2. Age: 16-70 years.
3. Patients with a diagnosis of advanced unresectable soft-tissue sarcoma and not candidates for surgical rescue including only the following subtypes: solitary fibrous tumor (SFT), synovial sarcoma, clear cell sarcoma, extraskeletal myxoid chondrosarcoma (EMC), alveolar soft part sarcoma and myxoid liposarcoma. Additionally, the Hospital Universitario Fundación Jiménez Díaz will include 2 desmoid tumor patients as proof of concept outside the total n.
4. Metastatic/locally advanced with recent progression (<6 months).
5. Patients should have received at least anthracyclines previously unless not indicated (SFT).
6. Measurable disease according to RECIST 1.1 criteria.
7. Patients must be willing to provide consent for the provision of mandatory biological samples for central pathology review (tumor sample from the three months prior to the start of treatment if the patient has not received any systemic therapy) and translational study (tumor blocks and blood).
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
9. Adequate hepatic, renal, cardiac, and hematologic function.
10. Laboratory tests as follows:

    * Absolute neutrophil count ≥1,500/mm³
    * Platelet count ≥100,000/mm³
    * Bilirubin ≤1.5 mg/dL
    * AST and ALT ≤2.5 times upper limit of normal
    * Creatinine ≤1.5 mg/dL
11. Left ventricular ejection fraction ≥50% by echocardiogram or MUGA scan.
12. Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to enrollment and agree to use birth control measures during study treatment and for 3 months after its completion. Patients must not be pregnant or nursing at study entry. Women/men of reproductive potential must have agreed to use a highly effective contraceptive method.
13. Subjects must be willing to avoid extensive sun exposure, phototherapy, and use of a tanning salon during trial participation.

Exclusion criteria:

Patients meeting any of the following exclusion criteria are not eligible to be enrolled in this study:

1. Previous treatment with CLK inhibitors.
2. Patients who have received any other anti-cancer therapy or investigational product in the last 28 days prior to enrollment.
3. Four or more systemic therapy lines for advanced disease.
4. Sarcoma subtypes other than the specified in the inclusion criteria.
5. Prior malignancy that required treatment or has shown evidence of recurrence (except for non-melanoma skin cancer, adequately treated cervical carcinoma in situ, superficial bladder carcinoma) during the 3 years prior to enrollment. Cancer treated with curative intent for >5 years previously and without evidence of recurrence will be allowed.
6. Any concurrent medical condition or disease (e.g., uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.) that is likely to interfere with study procedures.
7. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to Cycle 1 Day 1 (C1D1). Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
8. Pregnant or breastfeeding females.
9. Body surface area (BSA) <1.4 m2 at baseline, calculated by the Du Bois (33) or Mosteller (34) method.
10. Life expectancy of less than 3 months.
11. Major surgery within 28 days prior to C1D1.
12. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or dysfunction that could interfere with absorption of study treatment.
13. Inability or unwillingness to take supportive medications such as anti-nausea and anti anorexia agents as recommended by the NCCN CPGO for antiemesis and anorexia/cachexia (palliative care).
14. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
15. Subjects with a corrected QT interval (QTc) using Fridericia's formula (QTcF) > CTCAE v5.0 Grade 1 (>480 msec) based on the mean of triplicate evaluation at screening. In subjects with ventricular paced rhythm, a 50 msec subtraction should be applied to the QTc to calculate the QTcF, potential exceptions for subjects with pacemakers should be discussed with the Medical Monitor.
16. Subjects with clinically significant ventricular tachycardia (VT), atrial fibrillation (AF), ventricular fibrillation (VF), second or third degree heart block.
17. Subjects with myocardial infarction (MI) within 1 year, Class II-IV congestive heart failure (CHF) per New York Heart Association (NYHA) classification, or clinically significant coronary artery disease (CAD).
18. Subjects currently using or anticipating the need for food or drugs known to strongly inhibit or induce CYP3A4, such as ketoconazole, itraconazole, erythromycin, or rifampin, within 10 days prior to first dose of study medication.
19. Subjects with retinal abnormalities, specifically diabetic retinopathy, macular degeneration, other forms of retinal degenerative disease, or other retinal findings that may place the subject at risk (the latter should be discussed with the Medical Monitor).
20. Subjects with known active human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection.
21. Patient is unwilling to participate in the translational study (not providing mandatory written consent for tumor and blood samples).

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the progression-free survival rate (PFSR) at 3 months. | 3 months
  PFSR-3m (according to central radiology assessment): Efficacy measured by the PFSR at 3 months, which is defined as the percentage of patients who did not experience radiological progression according to RECIST v1.1 or death due to any cause since the date of treatment initiation until month 3 after date of treatment initiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Oncology Department, HU Fundación Jimenez Diaz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No